CLINICAL TRIAL: NCT01505335
Title: The Use of Novel us Device (Jetguide) to Measure the Distance to the Roof of the IAC (Inferior Alveolar Canal)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0460-11-RMB CTIL
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Comparison Between Ultrasound and Clinical Measurements
Keywords: alveolar nerve, inferior; ultrasound; digital radiography, dental; nerve injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Implant osteotomy measurements: Drilled implant locations
  Interventions: Device: US depth measurements

INTERVENTIONS:
Device: US depth measurements — Measurement of the distance between the apex of the drilled implant site and the IAC
  Other Names: Jetguide; Ultrasonic measurement device

SUMMARY:
The purpose of this human clinical trial is to validate the accuracy of Jetguide® US device in detecting the inferior alveolar canal (IAC) and to compare it to measurements performed on computerized tomography images.

DETAILED DESCRIPTION:
To date, the most accurate method to assess the distance from the alveolar crest to the IAC is cone beam computerized tomography (CBCT). This technique carries with it some potential concerns, including measurements errors, inability to perform intra-operative radiographs substantial financial and radiation costs.

In the present study patients will have a CBCT of the mandible taken. Sites where implants will be inserted will be marked on the CBCT, measurements of the distance from bone crest to the roof of the inferior alveolar canal (BC-IAC) will be performed.

During implant surgery the depth of the osteotomy (OD) will be measured using a periodontal probe; OD and the distance from the bottom of the osteotomy to the roof of the IAC (residual distance - RD) will be measured using a standard JetGuide® device. In addition, standard panoramic radiographs will be taken with a surgical gauge in the osteotomy which will enable us to measure the RD radiographically.

The correlation between the radiographic and clinical BC-IAC distance will be the primary outcome variable. The same correlation for the RD between the Jetguide readings and the linear measurements on the panoramic radiographs will serve as the secondary outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* missing teeth in the premolar and molar areas of the lower jaw

Exclusion Criteria:

* pregnancy
* pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects attentding the clinic, requiring dental implant therapy in the posterior part of the lower jaw.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Eli Machtei, Principal Investigator — Rambam Health Care Campus, Haifa, Israel
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel